CLINICAL TRIAL: NCT01692561
Title: Study Title: Brain Transmitters/Metabolites, Magnetic Resonance Spectroscopy, and Brain Connectivity: Diagnostic Strategies to Study the Effects of Non-Pharmacologic Therapies for Dysautonomia and Chronic Nausea
Brief Title: MRI to Assess the Effects of Dysautonomia and Chronic Nausea on Brain Transmitters
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: WFMCMRI 001; JEF MRI 001 (Other Grant/Funding Number: The Center for Biomolecular Imaging)
Record Dates: First submitted 2012-09-11; First posted 2012-09-25 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Dysautonomia
Keywords: Dysautonomia; Postural orthostatic tachycardic hypotension; Neurocardiogenic vasovagal syncope
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- normaL: Healthy subjects without symptoms of dysautonomia.
- Neurocardiogenic syncope: Fainting due to sudden drop in blood pressure.
- Orthostatic hypotension: Sudden decrease in blood pressure while standing.
- Postural Orthostatic Tachycardic Syndrome: Increased heart rate when standing.

SUMMARY:
The purpose of this research study is to better understand what causes dysautonomia and how this affects blood pressure and pulse. Dysautonomia is a condition of the autonomic nervous system. It is associated with fluctuations in blood pressure and pulse and may cause symptoms of nausea and belly pain, fatigue, excessive thirst, lightheadedness, dizziness, feelings of anxiety or panic, and fainting. A common example of dysautonomia is postural orthostatic tachycardia syndrome or POTS. Sometimes symptoms worsen when people move from lying down to standing, called orthostatic intolerance. We would like to learn more about the link between orthostatic intolerance and nausea. While medications currently used to treat orthostatic intolerance and nausea have proven to be effective in some patients, this may not be the best treatment for everyone as long term use could pose certain risks including high blood pressure. In order to provide a more focused and safer treatment for patients suffering from nausea and orthostatic intolerance, we have looked at how the blood pressure, pulse, and certain blood tests change during a tilt table test. This test helps to create the same circumstances that patients with orthostatic intolerance experience when they stand. To better understand if some of these problems are associated with the brain, we will study MRI in patients with dysautonomia compared to children without dysautonomia. This information may allow us to use alternative and safer treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have completed tilt autonomic testing
* subjects from 9 - 18 years of age

Exclusion Criteria:

* subjects who have a metabolic, mechanical, or mucosal inflammatory cause which has been defined to explain their gastrointestinal symptoms
* Patients with cardiac or cardiovascular disease, malignancy, psychiatric illness, neurodevelopmental delay, or other co-morbid conditions
* Patients with with pacemakers, implanted devices, or any other MRI contraindications will be excluded from this study.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A combination of male and female subjects who are healthy or ahve dysautonomia/
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-06-11 (Actual); Study Completion 2013-06-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the implication of dysautonomia on the brain and better evaluate its potential mechanistic process. | Assessments will occur in a one and a half hour visit.
  The first objective of the proposed project is to study central transmitter/metabolite profiles using in vivo 1H Magnetic Resonance Spectroscopy (MRS) in children with dysautonomia diagnosed by tilt table testing compared to healthy children without symptoms of dysautonomia. The second objective will be to determine whether dysautonomia associated with nausea and cardiovascular instability shares common alterations in brain networks. We will be using cognitive and sensory processing tasks based on our prior experience with both traditional fMRI and network analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Diz, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Fortunato JE, Laurienti PJ, Wagoner AL, Shaltout HA, Diz DI, Silfer JL, Burdette JH. Children with chronic nausea and orthostatic intolerance have unique brain network organization: A case-control trial. Neurogastroenterol Motil. 2022 Apr;34(4):e14271. doi: 10.1111/nmo.14271. Epub 2021 Oct 4. PMID 34606665